CLINICAL TRIAL: NCT06544109
Title: Venetoclax for Prevention of Differentiation Syndrom (DS) in Acute Promyelocytic Leukemia (APL) Patients : An Open-lable, Single-arm, Multicenter, Phase Ⅱ Clinical Trail
Brief Title: Venetoclax for Prevention of Differentiation Syndrom in Acute Promyelocytic Leukemia Patients
Acronym: Ven APL
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SZQ002
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-08

CONDITIONS: Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm Description:the Venatoclax regimen to prevent DS (Experimental): The patient with suspected APL should be treated with ATRA or Venetoclx depending on its WBC counts and rapid diagnosis of APL was made at the same time. Once APL was diagnosed, patients were initially treated with ATRA 25 mg/m2/d and ATO 0.16 mg/kg/d. During the induction regimen, patients in whom the WBC counts increased to more than 2 × 109/L received Venetoclax and DS was suspected received dexamethasone or ruxolitinib.
  Interventions: Drug: venetoclax

INTERVENTIONS:
Drug: venetoclax — patients in whom the WBC counts increased to more than 2 × 109/L received Venetoclax

SUMMARY:
This study is to assess the efficacy and safety of venetoclax for prevention of DS in APL patients undergoing ATRA/ATO induction regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent must have the ability to understand and be willing to participate in the study and sign the informed consent.
2. patients must have confirmation of APL by WHO criteria, previously untreated, and eligible for treatment with intensive chemotherapy as defined by the following: Cardiac history of congestive heart failure requiring treatment or ejection fraction ≤ 50% or chronic stable angina. Diffusing capacity of the lung for carbon monoxide (DLCO) ≤ 65% or forced expiratory volume during the first second (FEV1) ≤ 65%. Creatinine clearance < 45 mL/min. Moderate hepatic impairment with total bilirubin > 1.5 × ULN. Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy.

Exclusion Criteria:

1. Patient is ineligible for treatment with intensive chemotherapy
2. Patient with active infection not controlled, active bleeding from vital organs
3. Patient with history of clinically significant drug or alcohol abuse that would adversely affect evaluation in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
the rate of differential symdrom | the induction regimen (21 days to 28 days)
  DS, known as retinoic acid syndrome, is a severe complication of ATRA or ATO during the differentiation of promyelocytes. Signs of DS are presented as fever, weight gain, hypertension, dyspnoea, radiographic opacities, peripheral edema and acute renal failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Qiu huiying, Suzhou, Jiangsu, China